CLINICAL TRIAL: NCT06048783
Title: Feasibility and Preliminary Effects of a Spiritual Care Strategy on Psychological Disorders in Critically Ill Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 220111005
Record Dates: First submitted 2023-08-24; First posted 2023-09-21 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Psychological Disorder; Critical Illness
Keywords: Post traumatic stress disorder; Intensive Care; Critically ill patients; Spiritual Care
MeSH Terms: conditions — Mental Disorders; Critical Illness; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Program of systematic and periodic spiritual accompaniment and care (Experimental): A minimum of 3 sessions of spiritual accompaniment by trained volunteers, considering a 1:1 ratio (patient:companion). The topics that will be proposed during the sessions are: sense of suffering, uncertainty, death, life after life, ideas about healing, forgiveness and guilt, etc. In addition, the spiritual needs of the participants will be explored through an instrument specially designed for this purpose and culturally adapted in Chile (FICA). The spiritual accompaniment sessions will be implemented preferably at a distance, using zoom or video call.
  Interventions: Behavioral: Program of systematic and periodic spiritual accompaniment and care
- Standard Care (No Intervention): It correspond to spiritual care currently offered by the hospital. This consists of the possibility of being assisted by a Catholic priest or being contacted by pastors from Protestant churches.

INTERVENTIONS:
Behavioral: Program of systematic and periodic spiritual accompaniment and care — Systematic and periodic spiritual accompaniment and care
  Arms: Program of systematic and periodic spiritual accompaniment and care

SUMMARY:
Studies in hospitalized patients have shown that a large percentage of them consider religion or spirituality to be an important factor in enabling them to cope with a serious illness. Studies conducted in the ICU, have shown that spiritual care from a chaplain/priest is associated with increased satisfaction in family members of critically ill patients, however, the focus has traditionally been on offering support to family members and not to patients. Interventions for critically ill patients have mostly been implemented by chaplains or a member of the health care team, primarily nurses. Although these studies show promising results in terms of quality of life, they mostly reflect the perspective of the health teams and not that of the patients, they are not evaluated with standardized instruments and, in general, they are not standardized strategies.

Given that this will be one of the first studies with patients who received care in the ICU, it is proposed to conduct a pilot and feasibility study to gather lessons to implement a larger study. Studies of this type place greater emphasis on evaluating the feasibility of implementing the intervention and therefore this study will seek to: (1) evaluate the feasibility of implementing the intervention in a hospital setting, including participant recruitment procedures; (2) evaluate how the intervention, format and manner of implementation is received by participants; (3) preliminarily evaluate the impact on psychological symptomatology associated with PICS at the end of the intervention, at 3 and 6 months post-intervention.

Showing the impact of spiritual care on health outcomes of individuals, through studies such as this one, may contribute to a paradigm shift from a biomedical perspective to a holistic view of ICU patients. Although the technological and advanced life support offered by the ICU is essential for critical patients, but survival of a severe disease without a good quality of life makes it necessary to seek strategies to improve this problem, which undoubtedly requires a comprehensive approach to the person, through medical-physiological care and spiritual care.

DETAILED DESCRIPTION:
Many patients who survive a critical illness suffer physical, psychological and cognitive problems, negatively impacting their quality of life, which has been termed Post-ICU Syndrome (PICS). Some studies have reported a residual effect several months after discharge from the ICU, affecting people's quality of life and functionality. Among the psychological symptoms of PICS are described symptoms of depression, anxiety and post-traumatic stress disorder (PTSD). It is estimated that at least 50% of ICU survivors will present psychological symptoms of PICS at discharge and other studies report that a quarter of survivors present PTSD symptoms one year after discharge from the ICU.

Spirituality should be an essential element of health care, as it is part of the essence of being human. International accreditation associations and scientific societies suggest incorporating spiritual care into the usual standards of care. Studies of hospitalized patients have shown that a large percentage of patients consider religion or spirituality to be an important factor in enabling them to cope with serious illness. And although previous studies have shown that chaplain/priest care is associated with increased satisfaction in family members of critically ill patients, the focus has traditionally been on offering support to family members and not to patients. However, there is a growing recognition of the need for a comprehensive approach in health care to provide spiritual support to ICU patients that is evaluated and contributes to improving the quality of life of these individuals. On the other hand, showing the impact of spiritual care on health outcomes of individuals, through studies such as this one, can contribute to a paradigm shift from a biomedical perspective to a holistic view of ICU patients. The technological and advanced life support offered by the ICU is essential for critically ill patients, but the survival of a severe disease without a good quality of life makes it necessary to seek strategies to improve this problem, which undoubtedly requires a comprehensive approach to the person, through medical-physiological care and spiritual care.

The proposed design aims to evaluate the feasibility of implementing a spiritual accompaniment intervention for patients who received care in the ICU, and to begin to implement it during hospitalization. This will provide information regarding the feasibility of implementing an intervention of this type in this context, offering it during hospitalization and its remote implementation process, once the patient is discharged. Considering that these studies work with small samples, it is not necessary to estimate the sample calculation. However, in order to obtain some preliminary results of the effect of the intervention, a sample of 15 people per group will be recruited and followed up until 6 months after discharge, which will allow us to evaluate changes over time in PICS symptoms. It is proposed that the intervention will begin during hospitalization, so that it will have a preventive nature and help mitigate the impact of ICU hospitalization on the development of mental health symptoms in patients. Participants will be randomly assigned to groups and will be evaluated considering intention to treat. On the other hand, gathering the perspective of volunteers, patients and research support team will provide us with inputs to improve the intervention and the best way to implement it.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has had at least 72 hours of Invasive Mechanical Ventilation
* Patient currently in ICU
* Glasgow 15 at the moment of the screening

Exclusion Criteria:

* Patient who required mechanical ventilation in another episode of hospitalization in the 2 months before screening.
* Patients with primary neurological or neurosurgical disease.
* Presence of mental or intellectual disability prior to hospitalization or communication/language barriers.
* Pre-existing comorbidity with a life expectancy not exceeding 6 months (eg, metastatic cancer).
* Readmission to the ICU (patients can only be included if they are on their first ICU admission of the present hospitalization).
* No fixed address for follow-up.
* Patients with moderate to severe visual or hearing impairment.
* Early limitation of therapeutic effort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment | From recruitment to enrollment (i.e. up to 120 days)
  Proportion of eligible patients that are consented and enrolled in the trial
Attendance Rate | 2 weeks
  Proportion of participants who attend all three intervention sessions
Follow-up rate | 3 and 6 months post ICU discharge
  Proportion of patients who attend all follow-up assessment
Intervention Satisfaction Survey | 1-2 weeks and 3 months after the last session
  Satisfaction of the intervened group with the spiritual care will be assessed by a satisfaction survey.

SECONDARY OUTCOMES:
Intervention Satisfaction Survey | 1-2 weeks after the last session
  Volunteer satisfaction with the spiritual care and accompaniment intervention will be assessed by a satisfaction survey.
Post traumatic syndrome assessed by the Revised impact event scale (IES-R) | 3 and 6 months post ICU discharge
  The post traumatic syndrome will be evaluated thanks to the chilean version of the Revised impact event scale (IES-R) giving a score going from 0 to 88. This scale has a score from 0 to 88, defining a post-traumatic stress disorder with a score higher than 43.
Anxiety and depression symptoms assessed by Hospital Anxiety and Depression Scale (HADS) | 3 and 6 months post ICU discharge
  The HADS is a 14-item(1 - 4 points) measure designed to assess anxiety and depression symptoms in medical patients. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D). Scores higher than 11 on either scale indicate a definitive case.
Perceptions of patients, volunteers and research team about the intervention, its components, training and recommendations, and difficulties encountered | 2-3 weeks after the last session
  At the end of the study, three focus group will be held with the participants, volunteers and the research team. In the focus group, the same questions will be asked to all participants and the verbal answers to these questions will be recorded with voice recorders. Thematic analysis method will be used in the evaluation of the data.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Repetto, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Repetto P, Ruiz C, Rojas V, Olivares P, Bakker J, Alegria L. Spiritual care for prevention of psychological disorders in critically ill patients: study protocol of a feasibility randomised controlled pilot trial. BMJ Open. 2025 Apr 3;15(4):e084914. doi: 10.1136/bmjopen-2024-084914. PMID 40180407